CLINICAL TRIAL: NCT04671979
Title: Lactate Dehydrogenase, Bowel Necrosis and Mortality in Acute Mesenteric Ischemia: Retrospective Cross-Sectional
Brief Title: Serum Lactate in Acute Mesenteric Ischemia
Status: Completed | Type: Observational
Sponsor: Universidad del Rosario (Other)
Responsible Party: Principal Investigator, Andrés Isaza Restrepo, MD, MSc, Universidad del Rosario
Other Study IDs: DVO005-1-431-CEI969
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Mesenteric Ischemia
Keywords: Biomarker; L-Lactate; Mortality
MeSH Terms: conditions — Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lactate Dehydrogenase — All the patients that arrived at the hospital with symptoms of mesenteric ischemia, had a registered lactate dehydrogenase. We compared the value with the patient's outcomes.

SUMMARY:
Background: Acute mesenteric ischemia is a vascular emergency with high mortality because of ambiguous symptomatology and a lack of early diagnostic markers. Lactate dehydrogenase has been described as a mortality biomarker and bowel necrosis length too. Nevertheless, the association between them has been mildly studied. Our objective was to evaluate the association between serum lactate admission levels, bowel necrosis extension, and mortality. Additionally, we performed a mortality characterization.

Materials and Methods: A retrospective cross-sectional study was designed. We reviewed patients' clinical records with acute mesenteric ischemia that attended a hospital between 2012 and 2018. We compared serum lactate admission levels with bowel necrosis length and mortality. A receiver operating characteristic curve was performed on the last association. As post hoc analysis, a classification and regression tree on mortality was fitted.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Required urgent laparotomy with a postoperative diagnosis of acute mesenteric ischemia
* Attended the private academic hospital, between 2012 and 2018
* Had a registered serum lactate dehydrogenase at admission

Exclusion Criteria:

* Secondary causes of AMI
* Chronic intestinal ischemic
* Patient records with no description of the serum lactate dehydrogenase or extension of intestinal necrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seventy-four cases were identified that met the study's criteria. The patients' average age was 73.5 (SD, 10.7) years, and 44 (60%) were men. The mean body mass index was 25 (SD, 2.9) kg/m2. Fifteen (20%) of the patients presented non-occlusive acute mesenteric ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Serum Lactate in mmol/l | 30 days
Bowel necrosis length in cm | 30 days
Percentage of patients that died between 30 postsurgical days, % | 30 days

SECONDARY OUTCOMES:
Cut value of lactate levels as a predictor of mortality, in mmol/l | 30 days
  A receiver operating characteristics curve

CONTACTS AND LOCATIONS:
Locations (1):
- Andres Isaza Restrepo, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
We don't plan to share de IPD.